CLINICAL TRIAL: NCT02591888
Title: The Impact of Liposomal Bupivacaine Administered Following Placement of a Transobturator Suburethral Sling for Stress Urinary Incontinence: A Randomized Placebo-controlled Trial
Brief Title: Impact of Liposomal Bupivacaine Administered Following Placement of a Transobturator Suburethral Sling
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult to enroll; since a similar research project on a different population showed no significance the study has been closed.
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-081
Record Dates: First submitted 2015-02-26; First posted 2015-10-30 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal bupivacaine (Active Comparator): Subjects in this arm will received the drug - liposomal bupivacaine 30 ml.
  Interventions: Drug: Liposomal bupivacaine
- Placebo (Placebo Comparator): Subjects in this arm will received the placebo - normal saline 30 mL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — At the completion of the procedure, and at least 20 minutes after the injection of lidocaine with epinephrine (routine for the surgical procedure), those subjects in the placebo arm will have the 30ml of normal saline injected.
  Other Names: Normal Saline
  Arms: Placebo
Drug: Liposomal bupivacaine — At the completion of the procedure, and at least 20 minutes after the injection of lidocaine with epinephrine (routine for the surgical procedure), those subjects in the placebo arm will have the 30ml of dilutional liposomal bupivacaine injected.
  Other Names: Exparel
  Arms: Liposomal bupivacaine

SUMMARY:
Liposomal bupivacaine or placebo will be administered at the end of a transobturator midurethral sling to determine if there is a difference in a patient's perceived postoperative pain.

DETAILED DESCRIPTION:
The investigators aim to evaluate the use of liposomal bupivacaine to reduce postoperative pain from placement of transobturator slings for the treatment of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Planning for outpatient surgical treatment of SUI with placement of a transobturator suburethral sling under general anesthesia

Exclusion Criteria:

* Pregnant or nursing
* Allergy to bupivacaine
* History of drug/alcohol abuse
* Severe cardiovascular, hepatic, renal disease, or neurological impairment°
* Long-acting opioid within 3 days or any opioid use within 24 hours before surgery
* Contraindication to:
* acetaminophen
* oxycodone
* non-steroidal anti-inflammatory drugs (NSAID)
* Administration of an investigational drug within 30 days before study
* Chronic pain syndromes
* Daily NSAID/opioid use
* Patients having concomitant procedures or not undergoing general anesthesia
* Patients who require a concomitant anterior repair or urethrocele repair will not be excluded as this requires the same dissection in the anterior vaginal wall.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 4 hours after being discharged home
  To determine if liposomal bupivacaine administered at the completion of a transobturator suburethral sling will result in decreased postoperative pain compared to placebo.

SECONDARY OUTCOMES:
Likert scale to rate their level of satisfaction with their postoperative pain control. | At 1 and 2 weeks postoperatively
  To assess the amount of oral narcotic required for pain control following administration of liposomal bupivacaine or placebo at the completion of a transobturator sling procedure.

OTHER OUTCOMES:
VAS to rate their level of satisfaction with their postoperative pain control. | At 1 & 2 weeks postoperatively
  To assess the amount of oral narcotic required for pain control following administration of liposomal bupivacaine or placebo at the completion of a transobturator sling procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Catrina C Crisp, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No